CLINICAL TRIAL: NCT01850706
Title: Evaluation of Urinary Nerve Growth Factor as an Objective Tool to Assess Therapeutic Outcome in Patients With Detrusor Overactivity Undergoing Treatment With Sacral Neuromodulation
Brief Title: UNGF Assessment in Patients With Detrusor Overactivity Undergoing Sacral Neuromodulation
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Medtronics, Inc. (Industry)
Responsible Party: Principal Investigator, Dara Shalom, Principal Investigator, Northwell Health
Other Study IDs: 11-060A
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Detrusor Overactivity
Keywords: uNGF; urinary nerve growth factor; detrusor overactivity; InterStim; sacral neuromodulation; sacral nerve stimulation; quality of life; questionnaire; urodynamic detrusor overactivity; overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find a noninvasive test to help physicians diagnose detrusor overactivity (DO), to use this urine test to help diagnose bladder problems, determine if treatments are working, and determine if patients are good candidates for interventions like sacral neuromodulation/Interstim Therapy.

ELIGIBILITY:
Inclusion Criteria:

* for controls: age greater than or equal to 18; female gender, ability to provide informed consent and complete study requirements; subject has to be without urinary symptoms
* for cases: age greater than or equal to 18; female gender; ability to provide informed consent and complete study requirements; the subject should have symptoms of detrusor overactivity, including urinary frequency, urgency, or urge incontinence, for greater than or equal to 3 months; urodynamic diagnosis of detrusor overactivity; failed treatment with behavioral modification and anticholinergic medication

Exclusion Criteria:

* active urinary tract infection; currently undergoing hemodialysis or has severe renal impairment; bladder tumors; uncontrolled diabetes mellitus; post void residual greater than 100ml; history of use of anticholinergic treatment within past 21 days; history of urinary tract operation within 6 months prior to screening; heart failure; uncontrolled hypertension; severe neurological disease; history of botox usage within 1 year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects over 18 years of age will be screened for eligibility relative to patient inclusion and exclusion criteria. If eligible to enroll, the nature and purpose of this study will be explained to the subject with a witness present. The subject will review and sign the written Informed Consent Form indicating informed consent and voluntary participation in the study. A copy of the consent form including all risks and benefits to research subjects is attached as a separate document.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
uNGF level in patients with urodynamically proven DO at baseline versus normal controls | 1 year
Change in uNGF levels in patients with urodynamic DO at baseline and 5 days, 1 month, 3 months, and 12 months after treatment with Interstim | 1 year

SECONDARY OUTCOMES:
Change in quality of life questionnaire scores in patients with urodynamic DO at baseline and at 5 days, 1 month, 3 months, and 12 months after treatment with Interstim | 1 year
Correlation between uNGF levels and scores on validated quality of life questionnaires for urinary incontinence | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States